CLINICAL TRIAL: NCT02762981
Title: Phase 1/2 Study of CORT125134 in Combination With Nab-paclitaxel in Patients With Solid Tumors
Brief Title: Study to Evaluate Relacorilant (CORT125134) in Combination With Nab-paclitaxel in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORT125134-550
Record Dates: First submitted 2016-04-11; First posted 2016-05-05 (Estimated); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Solid Tumors
Keywords: CORT125134; nab-paclitaxel; Triple-Negative Breast Cancer; Ovarian Epithelial Cancer; GR Antagonist; Glucocorticoid Receptor Antagonist; Pancreatic Cancer; Solid Tumors; Relacorilant; Abraxane
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Ovarian Epithelial; Pancreatic Neoplasms | interventions — relacorilant; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relacorilant with nab-paclitaxel (Experimental): Participants will be treated with relacorilant in combination with nab-paclitaxel at escalating dose levels in either a Continuous-Dosing Regimen or an Intermittent-Dosing Regimen.
  Interventions: Drug: Relacorilant with nab-paclitaxel

INTERVENTIONS:
Drug: Relacorilant with nab-paclitaxel — Relacorilant is supplied as capsules for oral dosing. Nab-paclitaxel administered as an IV infusion.
  Other Names: Abraxane; Nanoparticle albumin-bound paclitaxel; CORT125134

SUMMARY:
The purpose of this study was to assess the safety of the combination of relacorilant (CORT125134), a novel glucocorticoid receptor (GR) antagonist, and nab- paclitaxel in participants with solid tumors and to determine the preliminary efficacy of the combination of relacorilant and nab-paclitaxel. The structure for the study was a single arm, non-randomized, open- label, multicenter trial with no control group.

DETAILED DESCRIPTION:
The study consisted of two segments to evaluate alternative dosing schedules of relacorilant administered at escalating dose levels. Segment I was to evaluate a continuous-dosing regimen and Segment II was to evaluate an intermittent-dosing regimen. Enrollment in Segment I and Segment II were mutually exclusive, and the two segments enrolled participants concurrently.

In Segment I continuous-dosing cohorts, participants received a single nab-paclitaxel lead-in infusion on Day 1 of Week -2 before Cycle 1, and oral relacorilant lead-in once-daily of Week -1 before Cycle 1. After the Data Review Committee review of data for 2 dose levels, the nab-paclitaxel lead-in was discontinued. The lead-in period was followed by oral relacorilant administered continuously once daily, in combination with nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle. Segment 1 enrolled a total of 64 participants.

In Segment II intermittent-dosing cohorts, participants received a single relacorilant lead-in dose on Day -1 before Cycle 1, followed by oral relacorilant, administered intermittently the day before, the day of, and the day after nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle. Segment II enrolled a total of 21 participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with advanced or metastatic solid tumors who have disease progression after treatment with available therapies and for whom nab-paclitaxel treatment is appropriate.
* Measurable or evaluable disease.
* Up to 3 prior cytotoxic chemotherapeutics regimens or myelosuppressive therapies in the advanced setting.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* For Part 2 Only: Platinum-resistant ovarian, fallopian tube, or primary peritoneal cancer, or Triple Negative Breast Cancer with measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in at least 1 lesion, that in the opinion of the Investigator is appropriate to treat with nab-paclitaxel.

Exclusion Criteria:

* Any major surgery within 4 weeks prior to the first dose of study drug.
* Some protocol specified treatments prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Corcept Therapeutics
Locations (4):
- United States (4):
  - 038, Scottsdale, Arizona
  - 014, San Francisco, California
  - 001, Chicago, Illinois
  - 013, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pivonello R, Munster PN, Terzolo M, Ferrigno R, Simeoli C, Puglisi S, Bali U, Moraitis AG. Glucocorticoid Receptor Antagonism Upregulates Somatostatin Receptor Subtype 2 Expression in ACTH-Producing Neuroendocrine Tumors: New Insight Based on the Selective Glucocorticoid Receptor Modulator Relacorilant. Front Endocrinol (Lausanne). 2022 Jan 4;12:793262. doi: 10.3389/fendo.2021.793262. eCollection 2021. PMID 35058882
- See also: A phase 1/2 study of relacorilant + nab-paclitaxel (nab-pac) in patients (pts) with solid tumors: The dose-finding phase — http://ascopubs.org/doi/abs/10.1200/JCO.2018.36.15_suppl.2554

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The starting population included all study participants.
Groups:
- Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen: Following lead-in, participants received relacorilant 100 mg, administered orally once daily, in combination with nab-paclitaxel 60 mg/m^2 infusions on Days 1, 8, and 15 of each 28-day cycle.
- Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen: Following lead-in, participants received relacorilant 100 mg, administered orally once daily, in combination with nab-paclitaxel 80 mg/m^2 infusions on Days 1, 8, and 15 of each 28-day cycle.
- Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen: Following lead-in, participants received relacorilant 150 mg, administered orally once daily, in combination with nab-paclitaxel 80 mg/m^2 infusions on Days 1, 8, and 15 of each 28-day cycle.
- Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen: Following lead-in, participants received relacorilant 150 mg, administered orally the day before, the day of, and the day after nab-paclitaxel 80 mg/m^2 infusions on Days 1, 8, and 15 of each 28-day cycle.
- Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen: Following lead-in, participants received relacorilant 200 mg, administered orally the day before, the day of, and the day after nab-paclitaxel 100 mg/m^2 infusions on Days 1, 8, and 15 of each 28-day cycle.
Period: Overall Study
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
Started | 17 | 40 | 7 | 16 | 5
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 40 | 7 | 16 | 5
Not completed — Adverse Event | 2 | 3 | 1 | 1 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1
Not completed — Disease progression | 11 | 23 | 4 | 10 | 1
Not completed — Enrolled not treated | 1 | 5 | 0 | 2 | 0
Not completed — Other | 2 | 3 | 1 | 0 | 0
Not completed — Missing | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of relacorilant. The Statistical Report specified summarization of Baseline Characteristic results by Segment I and Segment II.
Groups:
- Total: Total of all reporting groups
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen | Total
Number analyzed (Participants) | 14 | 34 | 6 | 14 | 5 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (10.60) | 60.6 (12.81) | 56.8 (18.51) | 59.6 (12.02) | 64.8 (10.21) | 59.7 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 20 | 4 | 14 | 3 | 50
  Male | 5 | 14 | 2 | 0 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 2 | 0 | 8
  Not Hispanic or Latino | 13 | 31 | 4 | 12 | 5 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 1 | 2 | 6
  White | 12 | 31 | 4 | 9 | 2 | 58
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 14 | 34 | 6 | 14 | 5 | 73

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity
Description: The Maximum Tolerated Dose and the development regimen of relacorilant with nab-paclitaxel was determined by the number of participants with dose-limiting toxicities as defined in the protocol.
Time Frame: Up to completion of Cycle 1 (up to 28 days)
Population: The dose-limiting toxicity evaluable population was participants who completed 1 cycle of treatment and assessment or received at least 1 dose of relacorilant and discontinued treatment before completing Cycle 1 due to toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
Number analyzed (Participants) | 10 | 23 | 4 | 11 | 3
Participants | 0 | 8 | 2 | 2 | 3

2. Secondary Outcome: Number of Participants With One or More Adverse Events Related to Treatment With Relacorilant
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Up to 28 days after the last dose of study drug (Segment I: up to approximately 2.5 years, Segment II: up to approximately 1.5 years)
Population: The safety population was all enrolled participants who received at least 1 dose of relacorilant.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
Number analyzed (Participants) | 14 | 34 | 6 | 14 | 5
Participants | 13 | 24 | 5 | 13 | 5

3. Other Pre Specified Outcome: Objective Response Rate
Description: Objective response rate is defined by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as best response of complete response (CR) or partial response (PR) from the start of relacorilant or nab-paclitaxel, whichever is earliest, across all time points during study observation period (including both confirmed and unconfirmed responses).
Time Frame: Up to 512 days
Population: All enrolled participants who received at least 1 dose of relacorilant. The Statistical Plan specified summarization of Objective Response Rate results by Segment I and Segment II.
Measure: Count of Participants; unit: Participants
Groups:
- Segment I: Continuous Dosing Regimens: Following lead-in, participants received oral relacorilant once daily, in combination with nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle.
- Segment II: Intermittent Dosing Regimens: Following lead-in, participants received oral relacorilant, administered the day before, the day of, and the day after nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle.
Arm/Group | Segment I: Continuous Dosing Regimens | Segment II: Intermittent Dosing Regimens
Number analyzed (Participants) | 54 | 19
Participants | 7 | 2

4. Other Pre Specified Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is defined as the participants who have achieved CR or PR (including both confirmed and unconfirmed responses), or stable disease for 16 weeks or greater.
Time Frame: Up to 512 days
Population: All enrolled participants who received at least 1 dose of relacorilant. The Statistical Plan specified summarization of Clinical Benefit Rate results by Segment I and Segment II.
Measure: Count of Participants; unit: Participants
Arm/Group | Segment I: Continuous Dosing Regimens | Segment II: Intermittent Dosing Regimens
Number analyzed (Participants) | 54 | 19
Participants | 13 | 6

5. Other Pre Specified Outcome: Duration of Response
Description: Duration of response (DOR) is defined as the date that criteria are met for CR or PR until the first date that progressive disease or death is objectively documented, whichever occurs first. Participants with no documentation of disease progression or death on-study are censored at the date of last available tumor assessment
Time Frame: From the time of response up to the last disease assessment (up to 512 days)
Population: All enrolled participants who received at least 1 dose of relacorilant. This outcome measure assessed participants with confirmed responses to treatment. The Statistical Plan specified summarization of Duration of Response results by Segment I and Segment II.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Segment I: Continuous Dosing Regimens | Segment II: Intermittent Dosing Regimens
Number analyzed (Participants) | 7 | 2
months | 9.7 [5.4 to 10.7] | NA [0.95 to NA] — Median and upper limit of 95% confidence interval was not estimable due to low number of participants with events.

6. Other Pre Specified Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from date of first dose of relacorilant or nab-paclitaxel, whichever is earliest, to the date of documented disease progression per RECIST v1.1 or death for any cause, whichever occurs first. Participants with no documentation of disease progression or death on-study are censored at the date of last available tumor assessment.
Time Frame: Up to 512 days
Population: All enrolled participants who received at least 1 dose of relacorilant. The Statistical Plan specified summarization of Progression-free Survival results by Segment I and Segment II.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Segment II: Intermittent Dosing Regimens: Following lead-in, participants received oral relacorilant the day before, the day of, and the day after nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle.
Arm/Group | Segment I: Continuous Dosing Regimens | Segment II: Intermittent Dosing Regimens
Number analyzed (Participants) | 54 | 19
Months | 2.8 [2.1 to 4.0] | 3.7 [2.9 to 16.2]

7. Other Pre Specified Outcome: Overall Survival
Description: Overall survival is defined as the time from date of the first dose of relacorilant or nab paclitaxel, whichever is earliest, to the date of death for any cause. Participants with no documentation of death on-study are censored at the date at which they are last known to be alive.
Time Frame: Up to 512 days
Population: All enrolled participants who received at least 1 dose of relacorilant. The Statistical Plan specified summarization of Overall Survival results by Segment I and Segment II.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Segment I: Continuous Dosing Regimens | Segment II: Intermittent Dosing Regimens
Number analyzed (Participants) | 54 | 19
Months | 8.3 [5.2 to 10.9] | 16.5 [8.5 to NA] — Upper limit of 95% confidence interval was not estimable due to low number of participants with event.

8. Other Pre Specified Outcome: Best Response Rate in Participants With Tumor Glucocorticoid Receptor (GR) Above or Below the Median Overall Level
Description: Best response is defined by RECIST v1.1 as the best response recorded from the date of the first dose of relacorilant or nab-paclitaxel, whichever is earliest, across all time points during study observation period (including both confirmed and unconfirmed responses).
Time Frame: Up to 512 days
Population: The population was all enrolled participants who received at least 1 dose of relacorilant and had tumor biopsy tissue assessed for GR. These data were planned to be summarized by GR H-score category: above or below the overall median value.
Measure: Count of Participants; unit: Participants
Groups:
- GR H-score Above the Overall Median: Participants from Segment I and Segment II who had above the overall median GR H-score at Baseline. Segment I: following lead-in, continuous dosing participants received oral relacorilant once daily, in combination with nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle. Segment II following lead-in, intermittent dosing participants received oral relacorilant the day before, the day of, and the day after nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle.
- GR H-score Below the Overall Median: Participants from Segment I and Segment II who had below the overall median GR H-score at Baseline. Segment I: following lead-in, continuous dosing participants received oral relacorilant once daily, in combination with nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle. Segment II: following lead-in, intermittent dosing participants received oral relacorilant the day before, the day of, and the day after nab-paclitaxel infusions on Days 1, 8, and 15 of each 28-day cycle.
Arm/Group | GR H-score Above the Overall Median | GR H-score Below the Overall Median
Number analyzed (Participants) | 16 | 16
Participants
  Complete response | 1 | 0
  Partial response | 3 | 1
  Stable disease | 7 | 7
  Progressive disease | 4 | 4
  Missing or not evaluable | 1 | 4

9. Other Pre Specified Outcome: Pharmacokinetics: Area Under the Concentration-time Curve From Zero to 24 Hours (AUC0-24) of Plasma Relacorilant
Time Frame: Segment I: before dosing and up to 24 hours after dosing on Cycle 1 Day 8; Segment II: before dosing and up to 24 hours after dosing on Cycle 1 Day 1
Population: The population analyzed was participants in the Safety Population with adequate pharmacokinetic data. One participant in the Segment II: relacorilant 150 mg + nab-paclitaxel 80 mg/m^2 intermittent dosing group had insufficient data to evaluate AUC0-24 for relacorilant.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
Number analyzed (Participants) | 10 | 27 | 4 | 14 | 4
ng*h/mL | 3380 (139) | 3780 (110) | 7480 (50.0) | 3300 (104) | 7440 (146)

10. Other Pre Specified Outcome: Pharmacokinetics: AUC0-24 of Plasma Nab-Paclitaxel
Time Frame: as for outcome 9
Population: The population analyzed was participants in the Safety Population with adequate pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
Number analyzed (Participants) | 10 | 27 | 4 | 15 | 4
ng*h/mL | 2290 (48.5) | 3580 (67.5) | 3380 (12.7) | 3440 (62.8) | 5910 (73.7)

11. Other Pre Specified Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Plasma Relacorilant
Time Frame: as for outcome 9
Population: The population analyzed was participants in the Safety Population with adequate pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
Number analyzed (Participants) | 10 | 27 | 4 | 15 | 4
ng/mL | 363 (100) | 423 (88.8) | 767 (47.4) | 546 (89.4) | 897 (55.2)

12. Other Pre Specified Outcome: Pharmacokinetics: Cmax of Plasma Nab-Paclitaxel
Time Frame: as for outcome 9
Population: The population analyzed was participants in the Safety Population with adequate pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
Number analyzed (Participants) | 10 | 27 | 4 | 15 | 4
ng/mL | 1810 (71.0) | 2660 (69.9) | 1560 (79.3) | 2600 (70.0) | 3070 (41.5)

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last dose of study drug (Segment I: up to approximately 2.5 years, Segment II: up to approximately 1.5 years)
Arm/Group | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen
All-Cause Mortality (participants affected / at risk) | 12/14 | 19/34 | 5/6 | 4/14 | 4/5
Serious Adverse Events (participants affected / at risk) | 6/14 | 18/34 | 5/6 | 8/14 | 3/5
Other Adverse Events (participants affected / at risk) | 13/14 | 31/34 | 6/6 | 14/14 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen (N=14) | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen (N=34) | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen (N=6) | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen (N=14) | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen (N=5)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Corneal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cerebral artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Segment I: Relacorilant 100 mg + Nab-paclitaxel 60 mg/m^2 Continuous Dosing Regimen (N=14) | Segment I: Relacorilant 100 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen (N=34) | Segment I: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Continuous Dosing Regimen (N=6) | Segment II: Relacorilant 150 mg + Nab-paclitaxel 80 mg/m^2 Intermittent Dosing Regimen (N=14) | Segment II: Relacorilant 200 mg + Nab-paclitaxel 100 mg/m^2 Intermittent Dosing Regimen (N=5)
Nausea (Gastrointestinal disorders) | 7 | 13 | 3 | 10 | 2
Vomiting (Gastrointestinal disorders) | 6 | 13 | 3 | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 12 | 2 | 9 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 1 | 6 | 1
Constipation (Gastrointestinal disorders) | 4 | 7 | 1 | 4 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 4 | 4 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Dysgeusia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Throat irritation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal stoma complication (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 16 | 6 | 8 | 4
Pyrexia (General disorders) | 1 | 6 | 2 | 1 | 1
Mucosal inflammation (General disorders) | 1 | 4 | 0 | 3 | 2
Oedema peripheral (General disorders) | 1 | 4 | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 1 | 1 | 1
Early satiety (General disorders) | 1 | 1 | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (General disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 8 | 2 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7 | 4 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 6 | 0 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 2 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 4 | 2 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0 | 2
Oedema pheripheral (Metabolism and nutrition disorders) | 0 | 4 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 7 | 3 | 6 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 9 | 3 | 4 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 4 | 4 | 7 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 5 | 4 | 7 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 9 | 3 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 7 | 5 | 3 | 3
Headache (Nervous system disorders) | 2 | 7 | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 3 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4 | 5 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 12 | 1 | 6 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 9 | 1 | 5 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 8 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 2 | 0
Candida infection (Infections and infestations) | 0 | 3 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 3 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 1 | 0
Disturbance in attention (Psychiatric disorders) | 1 | 2 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 2 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 3 | 1 | 1 | 0
Oedema peripheral (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 1 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 2 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1
Blister (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 1 | 0 | 0
Bloody discharge (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Corcept Therapeutics as the Sponsor, has a proprietary interest in this study. Authorship and manuscript composition will reflect joint cooperation between multiple Investigators and sites and Corcept personnel. Authorship will be established before the writing of the manuscript. As this study involves multiple centers, no individual publications will be allowed before completion of the final report of the multicenter study except as agreed with Corcept.

DOCUMENTS (2):
  • Study Protocol (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT02762981/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT02762981/SAP_001.pdf